CLINICAL TRIAL: NCT01749618
Title: Closing the Gap in Care in Seronegative Inflammatory Arthritis: From Identification to Implementation of Treating to Target: A Randomized Trial of Feedback, Education, and Behavioural Change
Brief Title: Closing the Gap in Care in Seronegative Inflammatory Arthritis
Acronym: Metrix II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pope Research Corporation (Industry)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Metrix II
Record Dates: First submitted 2012-11-06; First posted 2012-12-17 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: SpA; PsA
Keywords: Seronegative Inflammatory Arthritis; SpA; PsA; Randomized; Behavioural Change
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No education or feedback (No Intervention): Rheumatologists randomized to this treatment arm receive no additional education or feedback about their systematic assessments of patients
- Education and Feedback (Experimental): Rheumatologists randomized to receive education and feedback participate in six web conferences designed to improve their systematic assessments of their patients, and are given feedback about their performances
  Interventions: Behavioral: Education and Feedback

INTERVENTIONS:
Behavioral: Education and Feedback — Rheumatologists are rated on how systematically they assess their patients, and receive six sessions of university accredited education about systematic assessments of patients with seronegative arthritis.
  Arms: Education and Feedback

SUMMARY:
Rheumatologists treating patients with seronegative arthritis will be randomized to treat their patients to a target or to treat their patients under their usual standard of care. All physicians will perform an initial chart audit. Following the initial chart audit, all physicians in the treat-to-target group will receive accredited educational training. Six months after the initial chart audit, all physicians will perform a repeat audit to see if patients are assessed more systematically and treated to a target of low disease state.

ELIGIBILITY:
Inclusion Criteria:

* Canadian Rheumatologist

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Improvement of Systematic Assessments | November 2012 - November 2013
  Physicians in the Education and Feedback arm are assessed via a needs assessment to identify the care gaps for their patients with inflammatory arthritis. After the education and feedback, they complete a second chart audit and their improvements in assessments is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, MD, MPH, FRCPC, Principal Investigator — Pope Research Corp., St. Joseph's Health Care, Western University
Locations (9):
- Canada (9):
  - Dr. Vandana Ahluwalia, Brampton, Ontario
  - Dr. Sanjay Dixit, Burlington, Ontario
  - Dr Pauline Boulos, Hamilton, Ontario
  - Dr. Nikhil Chopra, London, Ontario
  - Dr Angela Montgomery, Mississauga, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario
  - The Medical Centre, Peterborough, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Dr. Arthur Karasik, Toronto, Ontario